CLINICAL TRIAL: NCT04508855
Title: Safety and Efficacy of Switching From Direct Oral Anticoagulants to Low Molecular Weight Heparin in Cancer Patients With Atrial Fibrillation During Antineoplastic Therapy
Brief Title: Management of Atrial Fibrillation in Patients With Cancer (MAFIC Study)
Acronym: MAFIC
Status: Withdrawn | Type: Observational
Why Stopped: Not enough participants
Sponsor: AHEPA University Hospital (Other)
Collaborators: Theagenio Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Thomas Zegkos, Resident in Cardiology, AHEPA University Hospital
Other Study IDs: MAFIC_2020
Record Dates: First submitted 2020-08-08; First posted 2020-08-11 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cancer; Atrial Fibrillation
Keywords: Cancer; Anticoagulation; Atrial fibrillation; Direct oral anticoagulants; low molecular weight heparin
MeSH Terms: conditions — Neoplasms; Atrial Fibrillation | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients with atrial fibrillation: All patients will be assigned to receive subcutaneous LMWH in therapeutic doses
  More specifically the regimens will be as follows:
  Tinzaparin 175 units/Kg once daily; Enoxaparin 1unit/kg twice daily; Fondaparinux <50 kg, 5 mg SC once daily, 50-100 kg, 7.5 mg SC once daily, >100 kg, 10 mg SC once daily; Bemiparin 115 IU/kg once daily; <50kg, 5000IU, 50-70kg, 7.500 IU, >70kg, 10000IU Nadroparin: Patients weighing 40 to 100 kg: SC, 171 anti-factor Xa IU per kg of body weight once a day; patients weighing over 100 kg will not receive nadroparin because a treatment dosage has not been established; Dalteparin: 200 units IU/kg SC daily for 30 days, then 150 units IU/Kg SC daily Dose adjustments will occur only in case of renal insufficiency according to the medicine's SPC The treatment with the LMWH will last at least during the period of active antineoplastic therapy of cancer patients
  Interventions: Drug: Low molecular weight heparin

INTERVENTIONS:
Drug: Low molecular weight heparin — Switch from direct oral anticoagulants to low molecular weight heparin

SUMMARY:
The primary objective is to assess the safety and efficacy of switching from direct oral anticoagulants to low molecular weight heparin in cancer patients during antineoplastic therapy

DETAILED DESCRIPTION:
This is a single-arm prospective observational study aiming to explore the safety and efficacy of switching from direct oral anticoagulants (DOAC) to low molecular weight heparin (LMWH) in cancer patients with atrial fibrillation (AF) during antineoplastic therapy or for a maximum time period of 6 months.

AF is the most common sustained arrhythmia; it affects 1.5% to 2% of the general population, and this prevalence increases to 10% at 80 years of age and to 18% at 85 years of age. Given the increasing occurrence of malignancies in the elderly and the coexistence of other conditions predisposing to AF in cancer patients, an association between those 2 conditions would be expected. A study including 24,125 patients estimated a prevalence of AF of 2.4% at the time of cancer diagnosis. A recent prospective study of 34,691 middle-aged women without AF or cancer at baseline showed that new-onset AF was a risk marker of subsequent diagnosis of cancer (HR 1.48, 95% CI 1.25 to 1.75; p <0.001).

Moreover, patients with cancer are at significantly higher risk of developing venous thromboembolism (VTE) which sometimes may precede the diagnosis of the malignancy. The risk is even higher when the patient is poorly mobilized or hospitalized. On the other hand, some anticancer therapies and especially the novel angiogenesis inhibitors are associated with increased thrombogenicity.

According to current Guidelines, DOACs are preferred over vitamin K antagonist (VKA) therapy and LMWH in both AF and VTE in the general population. However, in the presence of active cancer the administration of LMWH is advised for patients who are hospitalized for any reason and/or receiving chemotherapy, unless there is a high bleeding risk. LMWH has more favorable outcomes in cancer patients than VKAs, both in the setting of primary or secondary thromboembolic prophylaxis while extended anticoagulation (beyond the first 6 months) may be considered for an indefinite period or until the cancer is cured. This is possibly related with the fact that LMWH present antitumour and antimetastatic effects and confer an increased survival benefit. It should be noted that currently there is no conclusive evidence regarding the safety and efficacy of DOACs in cancer patients and the first results seem contradictory.

A number of recent studies with the use of DOACs in cancer-associated venous thromboembolism have demonstrated that these drugs are effective with similar rates of recurrent VTE but higher rates of major bleeding compared to LMWH. However, there are particular disadvantages, especially during the period of chemotherapy, such as interactions between these agents and anticancer therapies (eg, potential interactions between DOACs and azole-antimycotic agents), as well as unknown pharmacokinetics from chemotherapy-related vomiting.

Putting things together, many patients who are under a DOAC due to AF or previous VTE/pulmonary embolism (PE) may be diagnosed with cancer. Moreover, the risk of VTE is 6-fold higher on intravenous chemotherapy. For this reason, current clinical practice suggests that LMWH is continued during treatment with intravenous chemotherapy. However, data on the efficacy and safety of this common approach is lacking. This is important, especially in the setting of gastrointestinal tumors (especially gastric and pancreatic disease) which pose a high bleeding risk and especially during the chemotherapy active period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with cancer other than basal-cell or squamous-cell skin cancer which was objectively confirmed and are programmed for antineoplastic treatment
2. Subjects between 18 to 75 years of age at inclusion
3. Subjects must weigh at least 40 kg at inclusion
4. Subjects receiving direct oral anticoagulant treatment (rivaroxaban, dabigatran, apixaban, edoxaban) for prevention of stroke and systemic embolism in non-valvular atrial fibrillation

Exclusion Criteria:

1. Patients that have active or serious bleeding within the previous two weeks
2. Patients that have conditions associated with high bleeding risk (active peptic ulcer, recent neurosurgery
3. Patients with platelet count below 50000 per cubic millimeter
4. Patients who have contraindications to heparin (heparin-induced thrombocytopenia)
5. Patients with calculated creatinine clearance < 30 ml/min using the Cockcroft-Gault formula
6. Women who are pregnant
7. Life expectancy less than 6 months
8. Anticoagulation contraindications
9. Recent brain surgery within 6 months
10. Vascular surgery within 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with cancer and atrial fibrillation receiving direct oral anticoagulants and antineoplastic therapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Major bleeding | 6 months
  Death or a decrease in hemoglobin level of ≥ 2 g/dL over 24 hours or the need for transfusion of ≥ 2 units of packed red cells or clinically overt bleeding at critical site (eg, intracranial, retroperitoneal)
Clinical relevant bleeding | 6 months
  Bleeding that does not meet the criteria for major bleeding, however, it requires medical treatment or it affects the patient's daily activity

SECONDARY OUTCOMES:
Deep vein thrombosis or pulmonary embolism | 6 months
  t The first episode of symptomatic, documented deep vein thrombosis or pulmonary embolism
Thromboembolic stroke or systemic embolism | 6 months
  The first episode of symptomatic, documented thromboembolic stroke or systemic embolism

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - AHEPA University Hospital, Thessaloniki
  - Theagenio Cancer Hospital, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines (CPG). 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation. Developed with the special contribution of the European Heart Rhythm Association. Eur Heart J. 2012 Nov;33(21):2719-47. doi: 10.1093/eurheartj/ehs253. Epub 2012 Aug 24. No abstract available. PMID 22922413
- [Background] Hu YF, Liu CJ, Chang PM, Tsao HM, Lin YJ, Chang SL, Lo LW, Tuan TC, Li CH, Chao TF, Chung FP, Liao JN, Chen TJ, Chen SA. Incident thromboembolism and heart failure associated with new-onset atrial fibrillation in cancer patients. Int J Cardiol. 2013 May 10;165(2):355-7. doi: 10.1016/j.ijcard.2012.08.036. Epub 2012 Sep 16. No abstract available. PMID 22989607
- [Background] Lee AY, Levine MN, Baker RI, Bowden C, Kakkar AK, Prins M, Rickles FR, Julian JA, Haley S, Kovacs MJ, Gent M; Randomized Comparison of Low-Molecular-Weight Heparin versus Oral Anticoagulant Therapy for the Prevention of Recurrent Venous Thromboembolism in Patients with Cancer (CLOT) Investigators. Low-molecular-weight heparin versus a coumarin for the prevention of recurrent venous thromboembolism in patients with cancer. N Engl J Med. 2003 Jul 10;349(2):146-53. doi: 10.1056/NEJMoa025313. PMID 12853587
- [Background] Young AM, Marshall A, Thirlwall J, Chapman O, Lokare A, Hill C, Hale D, Dunn JA, Lyman GH, Hutchinson C, MacCallum P, Kakkar A, Hobbs FDR, Petrou S, Dale J, Poole CJ, Maraveyas A, Levine M. Comparison of an Oral Factor Xa Inhibitor With Low Molecular Weight Heparin in Patients With Cancer With Venous Thromboembolism: Results of a Randomized Trial (SELECT-D). J Clin Oncol. 2018 Jul 10;36(20):2017-2023. doi: 10.1200/JCO.2018.78.8034. Epub 2018 May 10. PMID 29746227
- [Background] Raskob GE, van Es N, Verhamme P, Carrier M, Di Nisio M, Garcia D, Grosso MA, Kakkar AK, Kovacs MJ, Mercuri MF, Meyer G, Segers A, Shi M, Wang TF, Yeo E, Zhang G, Zwicker JI, Weitz JI, Buller HR; Hokusai VTE Cancer Investigators. Edoxaban for the Treatment of Cancer-Associated Venous Thromboembolism. N Engl J Med. 2018 Feb 15;378(7):615-624. doi: 10.1056/NEJMoa1711948. Epub 2017 Dec 12. PMID 29231094